CLINICAL TRIAL: NCT03302572
Title: Effectiveness of a Brief Information About Advanced Directives in Primary Care: A Randomized Clinical Trial
Brief Title: Effectiveness Brief Information Advanced Directives Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15/101
Record Dates: First submitted 2017-09-18; First posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Primary Care; Advance Directives; Randomized Controlled Trial
Keywords: primary care; advance directives; randomized controlled trial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief information group (Experimental): Patients will be given brief information about the existence of advance directives after resolving the reason for the visit for which they had come. This information will not last more than 3 minutes and will not be repeated on successive visits within the recruitment period. Also, an informative triptych will be given to the patient so that he can read it at home. These leaflets have been made by the regional Department of Health. They will be advised that we can extend the information or help them to do the document in the near future if they want, we will inform that we would wait for the answer 3 months. In case of interest, they can leave their information in the User Service by specifying name, telephone number and reference doctor or ask for an appointment again.
  Interventions: Other: Brief information group
- Control group (No Intervention): Patients who fall into a control group will only be attended to their reason for visiting and will be asked for the necessary data to obtain the independent variables if they do not appear in their history. If the patient in this group wants the information, he will be excluded from the study because he "refuses to participate."

INTERVENTIONS:
Other: Brief information group — Patients will be given oral brief information about the existence of advance directives after resolving the reason for the visit for which they had come. This information will not last more than 3 minutes and will not be repeated on successive visits within the recruitment period. Also, an informative triptych will be given to the patient so that he can read it at home. These leaflets have been made by the regional Department of Health. They will be advised that we can extend the information or help them to do the document in the near future if they want, we will inform that we would wait for the answer 3 months. In case of interest, they can leave their information in the User Service by specifying name, telephone number and reference doctor or ask for an appointment again.
  Arms: Brief information group

SUMMARY:
The knowledge and completion of advanced directives (ADs) by the population is generally low. Primary care could develop a very important role to inform and assist in the preparation of this document because of its accessibility.

Objective: To evaluate the effectiveness of an oral brief information and a brochure administered in primary care to improve the proportion of ADs records.

Design: Randomized clinical trial. Ambit: 7 offices from a urban health center which serves about 25,000 users older than 18 years.

Material and methods It will be administered randomly triptych and oral brief information about the existence of advance directives for people over 18 to attend the appointment of their family doctor for any reason (intervention group). It will be given the possibility of more extensive information if they wish and collaboration will be offered for the advance directive according to patient preferences. The control group will not receive any information. Follow-up: 3 months. Variables will be: number of people interested in ADs, number of ADs made and demographic data (gender, age, education level, race, comorbidities, religion, testament) in both groups. Statistical analysis: multiple linear regression, Poisson and Cox as response analyzed, with the intervention/control group as the main variable adjusting for potential confounders. Bivariate comparison using Student t test or Mann-Whitney test (continuous variables) and chi-square or Fisher's exact test (categorical variables). 165 subjects were required in the control group and 165 in the intervention group.

Conclusion: positive results of this study will bring out the brief information managed by family physicians increases the number of ADs thus facilitating the right to autonomy of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old who go to their family doctor by appointment.

Exclusion Criteria:

* - Patients with language barrier
* Patients younger than 18 years (advanced directives not provided for by law)
* Patients with altered decision-making ability according to computerized clinical history by coding in health problems or mentioned in a clinical course of computerized medical history : cognitive impairment, dementia, mental retardation diagnosed. Although there are studies on attitudes towards advanced directives of people with early cognitive impairment (Minimental> 18), it was decided to discard because the intervention should be brief. The cited study also concludes that this type of patients prefer to delegate decisions to the family.
* Patients who come spontaneously to their family doctor.
* Patients who have already been recruited previously in the study. Patients who may visit by appointment only on more than one occasion will only participate once and subsequent visits for recruitment will be excluded. In addition, there will be no reinforcement of the study intervention in these visits.
* Patients who have already formalized the advanced directives.
* Patients who do not wish to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Interest in or performance of advance directives | In 3 months
  Proportion of people interested in or performance of Advance Directives in 3 months in the adult population. They will be obtained at the moment that the patient shows interest in the intervention of when they performance the Advance Directives, or if not, by asking by appointment or by telephone within 3 months of their recruitment

SECONDARY OUTCOMES:
Baseline characteristics of those who perform or are interested in Advanced Directives | In 3 months
  Evaluate the baseline characteristics of those who perform or are interested in Advanced Directives (whether they are in the control or intervention group).
Baseline characteristics of those performing Advanced directives in intervention group | In 3 months
  To assess the baseline characteristics of those performing the Advanced Directives and those not within the intervention group
Reasons to performance Advanced directives | In 3 months
  Evaluate the reasons why patients finally formalize the document by open question (will be categorized if there is a limited number of responses, otherwise the reasons will be described qualitatively).

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Rando, Principal Investigator — Institut Català de la Salut
Locations (1):
- Institu Català de la Salut, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
For confidentiality

DOCUMENTS (2):
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03302572/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT03302572/SAP_001.pdf